CLINICAL TRIAL: NCT02689128
Title: Postoperative Nausea and Vomiting: A Prospective Observational Study to Estimate the Incidence and Risk Factors Over One Year in a Tertiary Teaching Hospital
Brief Title: Postoperative Nausea and Vomiting: to Estimate the Incidence and Risk Factors in a Tertiary Teaching Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Other Study IDs: 269/14a/tk
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Anesthesia; postoperative; nausea; vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative nausea and vomiting (PONV) is a frequent complication of surgery and anesthesia.

The aim of this study is to estimate the incidence and the risk factors of PONV at Jordan University Hospital over one year period.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a frequent complication of surgery and anesthesia, in the literature it reaches up to 70% of the surgical patients and it occurs after local and general anesthesia with surgery.

Locally in Jordan there was no proper clinical study to estimate PONV among surgical patients, the aim of this study is to estimate the incidence and the risk factors of PONV at Jordan University Hospital over one year period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoes anesthesia and surgery.
* Patients who suffer from postoperative nausea and vomiting for 24 hours.

Exclusion Criteria:

* Patients who suffer from postoperative nausea and vomiting after 24 hours.
* Patients who undergoes Day-case surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergoes anesthesia and surgery and suffer from postoperative nausea and vomiting for 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Alghanem, FFARCS, Study Chair — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hambridge K. Assessing the risk of post-operative nausea and vomiting. Nurs Stand. 2013 Jan 2-8;27(18):35-43. doi: 10.7748/ns2013.01.27.18.35.c9486. PMID 23431652